CLINICAL TRIAL: NCT03886272
Title: Relative Bioavailability of Intended Commercial Formulations (iCF) of BI 730357 Versus BI 730357 Trial Formulation 1 and Bioavailability Comparison of Three Different iCF Batches Following Oral Administration in Healthy Subjects (an Open-label, Single-dose, Randomised, 2-way and 3-way Crossover Trial)
Brief Title: A Study in Healthy Men and Women to Test if Taking Different Formulations of BI 730357 Tablets Influences the Amount of BI 730357 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1407-0032; 2018-004421-91 (EudraCT Number)
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 730357 (Test) (Experimental)
  Interventions: Drug: BI 730357 (Test)
- BI 730357 (Reference) (Experimental)
  Interventions: Drug: BI 730357 (Reference)

INTERVENTIONS:
Drug: BI 730357 (Test) — tablet
  Arms: BI 730357 (Test)
Drug: BI 730357 (Reference) — tablet
  Arms: BI 730357 (Reference)

SUMMARY:
The main objective of Trial Parts 1 and 2 is to investigate the relative bioavailability of two tablet strengths (low dose and high dose) of the intended Commercial Formulation of BI 730357 (Test, T) versus with the corresponding tablet strengths of Trial Formulation 1 (Reference, R).

The main objective of Trial Part 3 is to investigate the relative bioavailability of two iCF side batches of BI 730357 with coarse milled Active pharmaceutical ingredient (API)(Test coarse milled, Tc) and unmilled API (Test unmilled, Tu), respectively, versus the final iCF batch of BI 730357 with regularly milled API (Reference, R).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), PR), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom:

    --- implants, injectables, combined oral or vaginal contraceptives, intrauterine device
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
* Surgically sterilised (including hysterectomy)
* Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of Follicle-stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including Blood pressure (BP), PR or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 12 g per day for females and 24 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Female subjects will not be allowed to participate, if any of the following apply:

  -- Positive pregnancy test, pregnancy, or plans to become pregnant within 30 days after study completion
* Lactation
* Male subjects with Woman of childbearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of first administration of trial medication until 30 days after the last administration of trial medication
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Ooi QX, Kristoffersson A, Korell J, Flack M, L Plan E, Weber B. Bounded integer model-based analysis of psoriasis area and severity index in patients with moderate-to-severe plaque psoriasis receiving BI 730357. CPT Pharmacometrics Syst Pharmacol. 2023 Jun;12(6):758-769. doi: 10.1002/psp4.12948. Epub 2023 May 1. PMID 36919398
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, single dose, randomized, 2-way and 3-way crossover trial in healthy subjects compared the relative bioavailability of intended commercial formulations (iCF) of BI 730357 to BI 730357 trial formulation 1 (TF1); and compared the bioavailability of different iCF batches (coarse-milled vs. unmilled vs. regularly milled).
Pre-assignment Details: Only subjects that met all the study inclusion and non of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue medication was allowed for all patients as required.
Groups:
- 50 mg BI 730357 iCF (T1) / 50 mg BI 730357 TF 1 (R1): 1 tablet of 50 milligram (mg) BI 730357 intended commercial formulations (iCF) final batch was administered as a single oral dose with 240 milliliter (mL) water as test treatment 1 (T1) after an overnight fast of at least 10 hours (h), followed by a wash-out phase of at least 10 days, followed by 1 tablet of 50 mg BI 730357 tablet formulation 1 (TF1), administered as a single oral dose with 240 mL water as reference treatment 1 (R1) after an overnight fast of at least 10h.
- 50 mg BI 730357 TF1 (R1) / 50 mg 730357 iCF (T1): 1 tablet of 50 milligram (mg) BI 730357 tablet formulation (TF1) was administered as a single oral dose with 240 milliliter (mL) water as reference treatment 1 (R1) after an overnight fast of at least 10 hours (h), followed by a wash-out phase of at least 10 days, followed by 1 tablet of 50 mg BI 730357 intended commercial formulations (iCF) final batch, administered as a single oral dose with 240 mL of water at test treatment 1 (T1) after an overnight fast of at least 10h.
- 200 mg BI 730357 iCF (T2) / 200 mg BI 730357 TF1 (R2): 2 tablets of 100 milligram (mg) BI 730357 intended commercial formulation (iCF) final batch were administered as a single oral dose with 240 milliliter (mL) water as test treatment 2 (T2) after an overnight fast of at least 10 hours (h), followed by a wash-out phase of at least 10 days, followed by 2 tablets of 100 mg BI 730357 tablet formulation 1 (TF1), administered as single oral dose with 240 mL water as reference treatment 2 (R2) after an overnight fast of at least 10h.
- 200 mg BI 730357 TF1 (R2)/ 200 mg BI 730357 iCF (T2): 2 tablets of 100 milligram (mg) BI 730357 tablet formulation 1 (TF1) were administered as a single oral dose with 240 milliliter (mL) of water as reference treatment 2 (R2) after an overnight fast of at least 10 hours (h), followed by a wash-out phase of at least 10 days, followed by 2 tablets of 100 mg BI 730357 intended commercial formulation (iCF) final batch, administered as a single oral dose with 240 mL water as test treatment 2 (T2) after an overnight fast of at least 10h.
- 100 mg BI 730357 Regularly Milled (R3)/ Coarse-milled (T3c)/ Unmilled (T3u): 1 tablet of 100 milligram (mg) BI 730357 intended commercial formulation (iCF) final batch regularly milled active pharmaceutical ingredient (API) was administered as a single oral dose with 240 milliliter (mL) water as reference treatment 3 (R3) after an overnight fast of at least 10 hours (h), followed by a wash-out phase of at least 10 days, followed by 1 tablet of 100 mg BI 730357 iCF side batch coarse-milled API, administered as a single oral dose with 240 mL water as test treatment 3c (T3c) after an overnight fast of at least 10 h, followed by a wash-out phase of at least 10 days, followed by 1 tablet of 100 mg BI 730357 iCF side batch unmilled API, administered as a single oral dose with 240 mL water as test treatment 3u (T3u) after an overnight fast of at least 10 h.
- 100 mg BI 730357 Coarse Milled (T3c) / Unmilled (T3u)/Regularly Milled (R3): 1 tablet of 100 milligram (mg) BI 730357 intended commercial formulation (iCF) side batch coarse-milled active pharmaceutical ingredient (API) was administered as a single oral dose with 240 milliliter (mL) water as test treatment 3c (T3c) after an overnight fast of at least 10 hours (h), followed by a wash-out phase of at least 10 days, followed by 1 tablet of 100 mg BI 730357 iCF side batch unmilled API, administered as a single oral dose with 240 mL water as test treatment 3u (T3u) after an overnight fast of at least 10 h, followed by a wash-out phase of at least 10 days, followed by 1 tablet of 100 mg BI 730357 iCF final batch regularly milled API, administered as a single oral dose with 240 mL water as reference treatment 3 (R3) after an overnight fast of at least 10 h.
- 100 mg BI 730357 Unmilled (T3u) /Regularly Milled (R3)/Coarse Milled (T3c): 1 tablet of 100 milligram (mg) BI 730357 intended commercial formulation (iCF) side batch unmilled active pharmaceutical ingredient (API) was administered as a single oral dose with 240 milliliter (mL) water as test treatment 3u (T3u) after an overnight fast of at least 10 hours (h), followed by a wash-out phase of at least 10 days, followed by 1 tablet of 100 mg BI 730357 iCF final batch regularly milled API, administered as a single dose with 240 mL water as reference treatment 3 (R3) after an overnight fast of at least 10 h, followed by a wash-out phase of at least 10 days, followed by 1 tablet of 100 mg BI 730357 iCF side batch coarse-milled API, administered as a single oral dose with 240 mL water as test treatment 3c (T3c) after an overnight fast of at least 10 h.
Period: Period 1
Arm/Group | 50 mg BI 730357 iCF (T1) / 50 mg BI 730357 TF 1 (R1) | 50 mg BI 730357 TF1 (R1) / 50 mg 730357 iCF (T1) | 200 mg BI 730357 iCF (T2) / 200 mg BI 730357 TF1 (R2) | 200 mg BI 730357 TF1 (R2)/ 200 mg BI 730357 iCF (T2) | 100 mg BI 730357 Regularly Milled (R3)/ Coarse-milled (T3c)/ Unmilled (T3u) | 100 mg BI 730357 Coarse Milled (T3c) / Unmilled (T3u)/Regularly Milled (R3) | 100 mg BI 730357 Unmilled (T3u) /Regularly Milled (R3)/Coarse Milled (T3c)
Started | 7 | 7 | 7 | 7 | 5 | 5 | 5
Completed | 7 | 7 | 7 | 7 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | 50 mg BI 730357 iCF (T1) / 50 mg BI 730357 TF 1 (R1) | 50 mg BI 730357 TF1 (R1) / 50 mg 730357 iCF (T1) | 200 mg BI 730357 iCF (T2) / 200 mg BI 730357 TF1 (R2) | 200 mg BI 730357 TF1 (R2)/ 200 mg BI 730357 iCF (T2) | 100 mg BI 730357 Regularly Milled (R3)/ Coarse-milled (T3c)/ Unmilled (T3u) | 100 mg BI 730357 Coarse Milled (T3c) / Unmilled (T3u)/Regularly Milled (R3) | 100 mg BI 730357 Unmilled (T3u) /Regularly Milled (R3)/Coarse Milled (T3c)
Started | 7 | 7 | 7 | 7 | 5 | 4 | 5
Completed | 7 | 7 | 7 | 7 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | 50 mg BI 730357 iCF (T1) / 50 mg BI 730357 TF 1 (R1) | 50 mg BI 730357 TF1 (R1) / 50 mg 730357 iCF (T1) | 200 mg BI 730357 iCF (T2) / 200 mg BI 730357 TF1 (R2) | 200 mg BI 730357 TF1 (R2)/ 200 mg BI 730357 iCF (T2) | 100 mg BI 730357 Regularly Milled (R3)/ Coarse-milled (T3c)/ Unmilled (T3u) | 100 mg BI 730357 Coarse Milled (T3c) / Unmilled (T3u)/Regularly Milled (R3) | 100 mg BI 730357 Unmilled (T3u) /Regularly Milled (R3)/Coarse Milled (T3c)
Started | 0 (This study arm is part of two-way cross over design. No third period exists in two way cross over.) | 0 (This study arm is part of two-way cross over design. No third period exists in two way cross over.) | 0 (This study arm is part of two-way cross over design.No third period exists in two way cross over.) | 0 (This study arm is part of two-way cross over design. No third period exists in two way cross over.) | 5 | 4 | 5
Completed | 0 | 0 | 0 | 0 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg BI 730357 iCF (T1) / 50 mg BI 730357 TF 1 (R1) | 50 mg BI 730357 TF1 (R1) / 50 mg 730357 iCF (T1) | 200 mg BI 730357 iCF (T2) / 200 mg BI 730357 TF1 (R2) | 200 mg BI 730357 TF1 (R2)/ 200 mg BI 730357 iCF (T2) | 100 mg BI 730357 Regularly Milled (R3)/ Coarse-milled (T3c)/ Unmilled (T3u) | 100 mg BI 730357 Coarse Milled (T3c) / Unmilled (T3u)/Regularly Milled (R3) | 100 mg BI 730357 Unmilled (T3u) /Regularly Milled (R3)/Coarse Milled (T3c) | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 5 | 5 | 5 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.4 (8.5) | 36.6 (9.5) | 35.0 (9.5) | 29.3 (4.6) | 39.2 (8.3) | 26.0 (7.0) | 29.6 (4.6) | 33.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 3 | 1 | 4 | 1 | 18
  Male | 5 | 5 | 2 | 4 | 4 | 1 | 4 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 6 | 7 | 7 | 7 | 4 | 5 | 5 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 7 | 7 | 7 | 5 | 5 | 5 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 730357 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 730357 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: Within 3 hours before and 0.5, 1, 1.5, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 34, 47, 71, 119 and 167 hours after drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): The PKS included all subjects in the treated set (TS) who provided at least 1 primary or secondary PK endpoint that was not excluded due to a protocol deviation or due to PK non-evaluability. It was sufficient for each subject to contribute only 1 PK parameter value for 1 period.
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomol*hours/Liter (nmol*h/L)
Groups:
- 50 mg BI 730357 iCF (T1): 1 tablet of 50 mg BI 730357 intended commercial formulation (iCF) final batch was administered as a single oral dose with 240 mL water after an overnight fast of at least 10 h, as test treatment 1 (T1).
- 50 mg BI 730357 TF1 (R1): 1 tablet of 50 mg BI 730357 tablet formulation 1 (TF1) was administered as a single oral dose with 240 mL water after an overnight fast of at least 10 h, as reference treatment 1 (R1).
- 200 mg BI 730357 iCF (T2): 2 tablets of 100 mg BI 730357 intended commercial formulations (iCF) final batch were administered as single oral dose with 240 mL water after an overnight fast of at least 10 h, as test treatment 2 (T2).
- 200 mg BI 730357 TF1 (R2): 2 tablets of 100 mg BI 730357 tablet formulation 1 were administered as a single oral dose with 240 mL water after an overnight fast of at least 10 h, as reference treatment 2 (R2).
- 100 mg BI 730357 iCF, Unmilled API (T3u): 1 tablet of 100 mg BI 730357 intended commercial formulation (iCF) side batch with unmilled active pharmaceutical ingredient (API) was administered as a single oral dose with 240 mL water after an overnight fast of at least 10 h, as test treatment 3u (T3u).
- 100 mg BI 730357 iCF, Coarse-milled API (T3c): 1 tablet of 100 mg BI 730357 intended commercial formulation (iCF) side batch with coarse-milled active pharmaceutical ingredient (API) was administered as a single oral dose with 240 mL water after an overnight fast of at least 10 h, as test treatment 3c (T3c).
- 100 mg BI 730357 iCF, Regularly Milled API (R3): 1 tablet of 100 mg BI 730357 intended commercial formulation (iCF) final batch was administered as a single oral dose with 240 mL water, after an overnight fast of at least 10 h, as reference treatment 3 (R3).
Arm/Group | 50 mg BI 730357 iCF (T1) | 50 mg BI 730357 TF1 (R1) | 200 mg BI 730357 iCF (T2) | 200 mg BI 730357 TF1 (R2) | 100 mg BI 730357 iCF, Unmilled API (T3u) | 100 mg BI 730357 iCF, Coarse-milled API (T3c) | 100 mg BI 730357 iCF, Regularly Milled API (R3)
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 15 | 14
nanomol*hours/Liter (nmol*h/L) | 5870.79 (NA) — Geometric Standard Error (gSE) = 1.08 | 5197.06 (NA) — Geometric Standard Error (gSE) = 1.08 | 19970.22 (NA) — Geometric Standard Error (gSE) = 1.09 | 17292.36 (NA) — Geometric Standard Error (gSE) = 1.09 | 5318.07 (NA) — Geometric Standard Error (gSE) = 1.10 | 9028.63 (NA) — Geometric Standard Error (gSE) = 1.10 | 11568.30 (NA) — Geometric Standard Error (gSE) = 1.10
Statistical Analysis 1: Comparison: 50 mg BI 730357 iCF (T1) vs 50 mg BI 730357 TF1 (R1); Relative bioavailability; Test type: Other; p = 0.0413, ANOVA — P-value for ratio outside 80% -125%; The model includes fixed effects for 'sequence', 'period', and 'treatment'. 'Subjects within sequences' is included as random effect; Adjusted Geometric Mean Ratio (T1/R1)[%] = 112.96, 90% CI 2-sided [102.70 to 124.26] — The Adjusted Geometric Mean is geometric mean adjusted by treatment. Ratio is calculated as: T1/R1. Intra-individual geometric coefficient of variation (gCV) = 14.2
Statistical Analysis 2: Comparison: 200 mg BI 730357 iCF (T2) vs 200 mg BI 730357 TF1 (R2); Relative bioavailability; Test type: Other; p = 0.0776, ANOVA — P-value for ratio outside 80% - 125%; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric Mean Ratio (T2/R2)[%] = 115.49, 90% CI 2-sided [105.23 to 126.74] — The Adjusted Geometric Mean is geometric mean adjusted by treatment. Ratio is calculated as T2/R2. Intra-individual geometric coefficient of variation (gCV) = 13.9
Statistical Analysis 3: Comparison: 100 mg BI 730357 iCF, Coarse-milled API (T3c) vs 100 mg BI 730357 iCF, Regularly Milled API (R3); Relative bioavailability; Test type: Other; p = 0.6443, ANOVA — P-value for ratio outside 80% - 125%; [statistical method as in outcome 1, analysis 1]; Adj. Geometric Mean Ratio (T3c/R3) [%] = 78.05, 90% CI 2-sided [69.71 to 87.38] — The Adjusted Geometric Mean is geometric mean adjusted by treatment. Ratio is calculated as Tc3/R3. Intra-individual geometric coefficient of variation (gCV) = 17.6
Statistical Analysis 4: Comparison: 100 mg BI 730357 iCF, Unmilled API (T3u) vs 100 mg BI 730357 iCF, Regularly Milled API (R3); Relative bioavailability; Test type: Other; p = 1.00, ANOVA — P-value for ratio outside 80% - 125%; [statistical method as in outcome 1, analysis 1]; Adj. Geometric Mean Ratio (T3u/R3) [%] = 45.97, 90% CI 2-sided [41.05 to 51.48] — The Adjusted Geometric Mean is geometric mean adjusted by treatment. Ratio is calculated as T3u/R3. Intra-individual geometric coefficient of variation (gCV) = 17.6

2. Primary Outcome: Maximum Measured Concentration of BI 730357 in Plasma (Cmax)
Description: Maximum measured concentration of BI 730357 in plasma (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanomol/Liter (nmol/L)
Arm/Group | 50 mg BI 730357 iCF (T1) | 50 mg BI 730357 TF1 (R1) | 200 mg BI 730357 iCF (T2) | 200 mg BI 730357 TF1 (R2) | 100 mg BI 730357 iCF, Unmilled API (T3u) | 100 mg BI 730357 iCF, Coarse-milled API (T3c) | 100 mg BI 730357 iCF, Regularly Milled API (R3)
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 15 | 14
nanomol/Liter (nmol/L) | 257.57 (NA) — Geometric Standard Error (gSE) = 1.07 | 178.10 (NA) — Geometric Standard Error (gSE) = 1.07 | 605.33 (NA) — Geometric Standard Error (gSE) = 1.06 | 466.75 (NA) — Geometric Standard Error (gSE) = 1.06 | 175.51 (NA) — Geometric Standard Error (gSE) = 1.09 | 317.95 (NA) — Geometric Standard Error (gSE) = 1.09 | 423.42 (NA) — Geometric Standard Error (gSE) = 1.09
Statistical Analysis 1: Comparison: 50 mg BI 730357 iCF (T1) vs 50 mg BI 730357 TF1 (R1); Relative bioavailability; Test type: Other; p = 0.9485, ANOVA — P-value for ratio outside 80% - 125%; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric Mean Ratio (T1/R1)[%] = 144.62, 90% CI 2-sided [124.82 to 167.57] — The Adjusted Geometric Mean is geometric mean adjusted by treatment. Ratio is calculated as T1/R1. Intra-individual geometric coefficient of variation (gCV) = 22.1
Statistical Analysis 2: Comparison: 200 mg BI 730357 iCF (T2) vs 200 mg BI 730357 TF1 (R2); Relative Bioavailability; Test type: Other; p = 0.7813, ANOVA — P-value for ratio outside 80% - 125%; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric Mean Ratio (T2/R2)[%] = 129.69, 90% CI 2-sided [119.51 to 140.73] — The adjusted geometric mean is geometric mean adjusted by treatment. Ratio is calculated as T2/R2. Intra-individual geometric coefficient of variation (gCV) = 12.2
Statistical Analysis 3: Comparison: 100 mg BI 730357 iCF, Coarse-milled API (T3c) vs 100 mg BI 730357 iCF, Regularly Milled API (R3); Relative Bioavailability; Test type: Other; p = 0.7616, ANOVA — P-value for ratio outside 80% - 125%; [statistical method as in outcome 1, analysis 1]; Adj. Geometric Mean Ratio (T3c/R3) [%] = 75.09, 90% CI 2-sided [64.58 to 87.32] — The Adjusted Geometric Mean is geometric mean adjusted by treatment. Ratio is calculated as = T3c/3. Intra-individual geometric coefficient of variation (gCV) = 23.5
Statistical Analysis 4: Comparison: 100 mg BI 730357 iCF, Unmilled API (T3u) vs 100 mg BI 730357 iCF, Regularly Milled API (R3); Relative Bioavailability; Test type: Other; p = 1.00, ANOVA — P-value for ratio outside 80% - 125%; [statistical method as in outcome 1, analysis 1]; Adj. Geometric Mean Ratio (T3u/R3) [%] = 41.45, 90% CI 2-sided [35.61 to 48.25] — The adjusted Geometric Mean is geometric mean adjusted by treatment. Ratio is calculated as = T3u/R3. Intra-individual geometric coefficient of variation = 23.5

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 730357 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 730357 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomol*hours/Liter (nmol*h/L)
Arm/Group | 50 mg BI 730357 iCF (T1) | 50 mg BI 730357 TF1 (R1) | 200 mg BI 730357 iCF (T2) | 200 mg BI 730357 TF1 (R2) | 100 mg BI 730357 iCF, Unmilled API (T3u) | 100 mg BI 730357 iCF, Coarse-milled API (T3c) | 100 mg BI 730357 iCF, Regularly Milled API (R3)
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 15 | 14
nanomol*hours/Liter (nmol*h/L) | 6222.62 (NA) — Geometric Standard Error = 1.08 | 5600.47 (NA) — Geometric Standard Error = 1.08 | 21074.02 (NA) — Geometric Standard Error = 1.11 | 18464.52 (NA) — Geometric Standard Error = 1.11 | 5843.68 (NA) — Geometric Standard Error = 1.10 | 9585.79 (NA) — Geometric Standard Error = 1.09 | 11967.75 (NA) — Geometric Standard Error = 1.10
Statistical Analysis 1: Comparison: 50 mg BI 730357 iCF (T1) vs 50 mg BI 730357 TF1 (R1); Relative Bioavailability; Test type: Other; p = 0.0092, ANOVA — P-value for ratio outside 80% - 125%; The model included fixed effects for 'sequence', 'period', and 'treatment'. 'Subjects within sequences' is included as random effect; Adjusted Geometric Mean Ratio (T1/R1)[%] = 111.11, 90% CI 2-sided [102.87 to 120.01], Standard Deviation 11.5 — The Adjusted Geometric Mean is geometric mean adjusted by treatment. Ratio is calculated as T1/R1. Intra-individual geometric coefficient of variation (gCV) = 17.6
Statistical Analysis 2: Comparison: 200 mg BI 730357 iCF (T2) vs 200 mg BI 730357 TF1 (R2); Relative Bioavailability; Test type: Other; p = 0.0442, ANOVA — P-value for ratio outside 80% - 125%; [statistical method as in outcome 3, analysis 1]; Adjusted Geometric Mean Ratio (T2/R2)[%] = 114.13, 90% CI 2-sided [104.58 to 124.56] — The Adjusted Geometric Mean is geometric mean adjusted by treatment. Ratio is calculated as = T2/R2. Intra-individual geometric coefficient of variation (gCV) = 13.0
Statistical Analysis 3: Comparison: 100 mg BI 730357 iCF, Coarse-milled API (T3c) vs 100 mg BI 730357 iCF, Regularly Milled API (R3); Relative Bioavailability; Test type: Other; p = 0.4928, ANOVA — P-value for ratio outside 80% - 125%; [statistical method as in outcome 3, analysis 1]; Adj. Geometric Mean Ratio (T3c/R3) [%] = 80.10, 90% CI 2-sided [71.54 to 89.68] — The Adjusted Geometric Mean is geometric mean adjusted by treatment. Ratio is calculated as = T3c/R3. Intra-individual geometric coefficient of variation (gCV) = 17.6
Statistical Analysis 4: Comparison: 100 mg BI 730357 iCF, Unmilled API (T3u) vs 100 mg BI 730357 iCF, Regularly Milled API (R3); Relative Bioavailability; Test type: Other; p = 1.00, ANOVA — P-value for ratio outside 80% - 125%; [statistical method as in outcome 3, analysis 1]; Adj. Geometric Mean Ratio (T3u/R3) [%] = 48.83, 90% CI 2-sided [43.60 to 54.69] — [estimate comment as in outcome 1, analysis 4]

ADVERSE EVENTS:
Time Frame: [Serious and other adverse events]:Up to 7 days after drug administration. All-cause mortality was collected up to 16 days.
Description: Adverse events are reported on the treated set (TS). The TS included all subjects who were randomized and treated with at least 1 dose of trial drug.
Arm/Group | 50 mg BI 730357 iCF (T1) | 50 mg BI 730357 TF1 (R1) | 200 mg BI 730357 iCF (T2) | 200 mg BI 730357 TF1 (R2) | 100 mg BI 730357 iCF, Unmilled API (T3u) | 100 mg BI 730357 iCF, Coarse-milled API (T3c) | 100 mg BI 730357 iCF, Regularly Milled API (R3)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 3/14 | 4/14 | 7/14 | 8/14 | 2/14 | 3/15 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg BI 730357 iCF (T1) (N=14) | 50 mg BI 730357 TF1 (R1) (N=14) | 200 mg BI 730357 iCF (T2) (N=14) | 200 mg BI 730357 TF1 (R2) (N=14) | 100 mg BI 730357 iCF, Unmilled API (T3u) (N=14) | 100 mg BI 730357 iCF, Coarse-milled API (T3c) (N=15) | 100 mg BI 730357 iCF, Regularly Milled API (R3) (N=14)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 3 | 6 | 8 | 0 | 2 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT03886272/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT03886272/SAP_001.pdf